## The Evaluation Of The Efficiency Of Micro-osteoperforation

Date : April 28, 2016

Statistical Analysis Plan (SAP)

Data were analyzed by IBM SPSS (version: 25.0, IBM Corp., Armonk, New York, USA) statistical package program. Descriptive statistical data were number of units (n), percentage (%), mean  $\pm$  standard deviation ( $\bar{x} \pm$ ).

Correlation between the measurements (method error) was evaluated with intraclass correlation coefficient. In the assessment of the compatibility of the Model and Little perpendicularity index measurements, the intraclass correlation coefficient was specified with a 95% confidence interval.

The normal distribution of the numerical variables was evaluated by Shapiro-Wilks normality test and Q-Q graphs. Independent samples t test was used to compare the means between two independent groups of continuous measurements, and dependent sample t test was used to compare two dependent groups. Gender distribution between groups was evaluated using chi-square test.

The comparison of the groups according to time was made by means of two-way analysis of variance and generalized linear models in repeated measurements. Bonferroni test was used as multiple comparison test. The level of statistical significance was set at  $p \le 0.05$ .